CLINICAL TRIAL: NCT02652520
Title: Evaluation of a Marine OXYgen Carrier: HEMO2Life® for hypOthermic Kidney Graft Preservation, Before Transplantation
Brief Title: Evaluation of a Marine OXYgen Carrier: HEMO2Life® for hypOthermic Kidney Graft Preservation, Before Transplantation (OXYOP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OXYOP (RB 14.208)
Record Dates: First submitted 2015-12-22; First posted 2016-01-12 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: End Stage Renal Diseases
Keywords: Kidney transplantation; Organ preservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kidney transplantation (Experimental): HEMO2Life® use in organ preservation solution. Grafts removed and transplanted locally within the 6 kidney transplant centers participating in the study will be preserved with Hemo2life.
  Interventions: Procedure: HEMO2Life® use in organ preservation solution

INTERVENTIONS:
Procedure: HEMO2Life® use in organ preservation solution — The surgeon decides whether the local transplant kidney may be part of the study and whether it should be stored in static cold storage or machine perfusion. The transplant kidney will be perfused in situ before procurement with the Belzer UW® cold storage solution furnish by the BridgetoLife company. HEMO2Life® will then be added to preservation solution.

SUMMARY:
Kidney transplantation is the treatment of choice for end stage renal diseases, increasing life expectancy and quality of life. Improvement in organ preservation is a critical issue in this context.

This is a safety study evaluating the use of an oxygen carrier HEMO2Life® as an additive in organ preservation solution in kidney transplantation.

DETAILED DESCRIPTION:
Security of the use of HEMO2Life® will be analyzed by collecting all events within the first 3 months in terms of :

1. HEMO2Life® adverse effects
2. graft safety
3. recipient safety (any adverse event) Accountability search will be achieved for each of these events.

ELIGIBILITY:
Inclusion Criteria:

For Kidney :

The first ten local kidneys in each participating centers that do not meet the exclusion criteria.

* Graft retrieved in an adult donor
* Graft from a deceased donor after brain death (DBD)
* Graft locally transplanted in one of the 6 kidney transplant centers participating in the study
* Graft stored in preservation solution containing HEMO2Life®

For Patient :

Patient who signed an inform consent form In case of patient unable to signed an inform consent form for patient under judicial protection (supervision, guardianship) the inform consent form will be obtain from the patient himself and from the supervisor/guardianshiper/parents, they will signed together the patient inform consent form.

The probability of the inclusion of a patient unable to signed an inform consent form is low but we can't know the receiver before conditioning the graft.

Patient > 18 years old

Exclusion Criteria:

* Graft from a living donor
* Graft from a donor after cardiovascular death (DCD)
* Graft dedicated to a multi-organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
HEMO2Life® adverse effects | During 3 months
  All incidents and events of interest occurring during the use of HEMO2Life® will be collected
Graft safety | During 3 months
  Collecting any complication with particular attention to mascroscopic aspect, contamination of the conservation solution, surgical difficulties and thrombosis, primary non function, delayed graft function, slow recovery of graft function, acute rejection, or any other graft complications.
Recipient safety (any adverse event) | During 3 months
  All adverse events, even unrelated to HEMO2Life®, occuring during the first 3 months after transplantation will be collected. Vital signs and laboratory evaluations will be collected at D0, D1, D3, D7, D14, M1, M2 and M3 to evaluate the recipient safety

SECONDARY OUTCOMES:
Comparison of the graft survival criteria with a control population | Baseline to 12 months
  Results will be compared with patients from a case control group of grafts transplanted at the same time in the 4 transplant centers from the Spiesser group (Tours, Poitiers, Brest, Limoges). Groups will be formed after matching on sex, age and cold ischemia time thanks to the Astre database regrouping the data of all the transplant teams from the Spiesser group.
Histological evaluation of the graft on biopsies | pre-implantation to 3-month biopsies
  All biopsies are interpreted locally and classified according to the Banff classification. Interstitial fibrosis quantification using automated quantitative image analysis of biopsies will also be performed from each biopsy.
Analysis of markers involved in kydney regeneration and neovascularization and markers of cellular stress. | Baseline to 12 months
  Analysis of blood and urine biomarkers at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Yannick LE MEUR, Principal Investigator — Principal Investigator and Nephrology coordinator; Benoit BARROU, Principal Investigator — Urology coordinator
Locations (6):
- France (6):
  - CHRU Brest, Brest
  - CHU Limoges, Limoges
  - Hôpital Edouard Herriot, Lyon
  - Hôpital la Pitié Salpetrière, Paris
  - CHU Poitiers, Poitiers
  - CHRU de Tours, Tours